CLINICAL TRIAL: NCT06354751
Title: Maternity Care Experiences of Asylum-seeking and Refugee Women in Scotland
Acronym: MACAWS
Status: Recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 327236
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Refugee; Asylum-seeking Women; Maternity
Keywords: maternity care; Scotland; experiences

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The International Organisation of Migration reports that over half (52.4%) of international migrants in Europe are women. Evidence suggests that women with immigrant backgrounds often struggle to access healthcare across the world. Among migrant women, asylum-seeking and refugee women face higher risks of poor pregnancy and birth outcomes, including babies with low birth weight, physical and/or mental health problems or death related to pregnancy and/or childbirth. Previous studies have focused on immigrant women's experiences of care during pregnancy and birth and did not differentiate between asylum seekers, refugees, and economic migrants. This can make it difficult to compare studies accurately. This study focuses on asylum-seeking and refugee women, using the definitions provided by the United Nations. Asylum-seeking women refer to women who seek protection in a country other than their own and are waiting for a decision on their status. Asylum seekers become refugees once their application has been processed and accepted.

A scoping review was conducted to understand the experiences of asylum-seeking and refugee women accessing maternity care in the United Kingdom( UK), focusing on Scotland. The review found that all studies that focused on the experiences of asylum-seeking and refugee women accessing maternity care were mainly based in England. The review identified the presence of specialist migrant services in maternity settings in Scotland and across the UK. Still, there was no information on their implementation or impact on women's outcomes. Additionally, there is limited evidence in the UK on the perceptions of healthcare professionals providing care to asylum-seeking and refugee women.

This study aims to close this gap in research by exploring this area more deeply in Scotland through mixed-methods studies of surveys with asylum-seeking and refugee women and interviews with maternity care leaders, policymakers, maternity healthcare professionals, and asylum-seeking and refugee women.

DETAILED DESCRIPTION:
This study aims to understand how asylum-seeking and refugee women in Scotland experience maternity care and how healthcare professionals perceive working with asylum-seeking and refugee women in maternity services. To achieve this, the study will use an explanatory sequential design. This means that the study will begin with a survey, followed by interviews with selected participants, with the aim of explaining the survey results. More details about the study design are below.

Asylum-seeking and refugee women in Scotland will be invited to complete a survey online or on paper. This survey will ask questions about their experiences of using maternity services in Scotland, and women will have a chance to write comments or feedback if they wish. The survey should take no longer than 10-15 minutes to complete. Agreeing to join the study does not mean that the participants have to complete it, they are free to withdraw at any time before submission.

After that, in the interview study phase, asylum-seeking and refugee women in Scotland, including those who completed the survey and expressed interest in participating in the interview study, will be invited to participate in the interviews. Also, HealthCare Professionals (HCPs) will be invited to participate in interviews to talk about their experiences providing care to asylum-seeking and refugee women in Scotland. The interviews will last approximately 30-60 minutes. The interviews will help to gain an in-depth understanding of the survey results. Potential participants will be encouraged not to agree to participate in this research until they have answers to any questions. For in-person interviews, participants will be asked to sign a consent form to show they agreed to participate while verbal consent will be obtained for online interviews. The participants can withdraw at any time, without giving a reason. If the participant agrees to participate, they will be invited to participate in an interview with the researcher. The interview can be conducted either online or face-to-face. All interviews will be recorded using a password-protected audio recorder. The researcher will arrange a convenient time at a location of the participant's choice to participate in the interview. The participants will be reassured that there are no right or wrong answers and that they do not have to answer all the questions. They can ask the researcher to move on to the next question if they do not wish.

Statistical Package for Social Sciences (SPSS) statistical software will be used to conduct statistical analyses. Descriptive statistics and data visualisation will be employed to analyse quantitative data obtained from the survey. Free-text responses from the survey will be analysed using a thematic analysis approach. Any question in the survey without an answer will be considered a missing data point and will not be included in any analysis containing that variable.

The collected qualitative data from interviews will be entered into NVivo for coding, and inductive thematic analysis will be used, following Braun and Clarke's method. The mixed methods will enable the integration of quantitative and qualitative results during the interpretations and explanations. The findings will help inform local and national models of care and approaches and attitudes needed to support these women ultimately.

ELIGIBILITY:
( Phase one: Survey)

- Inclusion Criteria:

* Women aged 16 and over.
* Women who are or were or had been pregnant within the last 5 years.
* Women who were living in Scotland within the last 5 years and used National Health Service (NHS) maternity services.
* Asylum-seeking woman at the time of being pregnant or Refugee woman at the time of being pregnant.
* Able to understand written or spoken English, Arabic, Persian or Urdu sufficiently to complete the survey.

Exclusion Criteria :

* Women who are economic migrants or illegal migrants or hold British citizenship at the time of being pregnant and using maternity services within last five years in Scotland.
* Women who are asylum-seeking or refugee women and live in England or Wales or Northern Ireland.
* Women with insufficient English, Arabic, Persian or Urdu to participate in the online survey.

(Second phase: interview)

Inclusion Criteria for women:

* Women aged 16 and over.
* Women who can provide verbal or written consent.
* Women who are currently pregnant or have been pregnant within the last 5 years.
* Women who were living in Scotland within the last 5 years and used NHS maternity services.
* Asylum-seeking woman at the time of being pregnant or Refugee woman at the time of being pregnant.
* Able to understand written or spoken English or Arabic sufficiently to participate in the interview.

Exclusion Criteria for women:

* Women who are economic migrants or illegal migrants or hold/held British citizenship at the time of being pregnant and used maternity services within last five years in Scotland.
* Women who are asylum-seeking or refugee women and live in England, Wales or Northern Ireland.
* Women with insufficient English or Arabic to participate in the interviews.

Inclusion Criteria for HCPs:

* Currently employed in NHS Scotland in maternity services, including:

  * health care support worker,
  * midwife,
  * doctor and obstetrician,
  * Maternity care leader/manager.
* Able to provide verbal or written consent.

Exclusion Criteria for HCPs:

• HCPs working in other specialists (outside of the previously mentioned professions).

Ages: 16 Years to 50 Years | Sex: Female
Age Groups: Child, Adult
Study Population: The study population for the survey consists of asylum-seeking and refugee women who were pregnant or who had been pregnant in Scotland the last five years, regardless of the outcome of pregnancy ( e.g live birth, stillbirth, miscarriage or abortion).
  The study population for the interviews consists of two samples. First, asylum-seeking and refugee women who are pregnant or who had been pregnant in Scotland in the last five years, regardless of the outcome of pregnancy (e.g live birth, stillbirth, miscarriage or abortion). Second, the HCPs who are providing care to those women in maternity services in Scotland.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Exploring and understanding asylum-seeking and refugee women's experiences of maternity care in Scotland. | by May 2025
  A survey will be conducted to assess asylum-seeking and refugee women's experiences of maternity care in Scotland. This will be followed by a qualitative phase, during which semi-structured interviews with asylum-seeking and refugee women will provide an in-depth understanding of the findings of the survey.
Evidence of HCP's experiences of providing maternity care for asylum-seeking and refugee women in Scotland. | by May 2025
  In depth semi-structured interviews will be offered to HCPs to explore their experiences of providing care to asylum seeking and refugee women in maternity services in Scotland.

SECONDARY OUTCOMES:
Identification of the successful components of specialist migrant maternity services in Scotland. | by May 2025
  The results from the survey and interviews will help identify the specialist migrant maternity services in Scotland.
Identification of gaps between care pathways and practice (implementation gap) and how this affects the quality of maternity care and women's experiences of maternity services | by May 2025
  The mixed method analysis of the findings will help identify gaps between current care pathways and collected data from women's experiences of using maternity services in Scotland.
Information for policymakers on approaches needed to improve maternity care for refugee and asylum-seeking women at local and national levels. | by May 2025
  The findings of the study and its recommendations will be shared with maternity managers and policy makers to enhance women's experiences of maternity services and meet their needs in Scotland.

CONTACTS AND LOCATIONS:
Overall Officials: Mairead Black, PhD, Principal Investigator — UoA Reader
Locations (1):
- NHS Grampian, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No